CLINICAL TRIAL: NCT00965250
Title: Multicenter Phase II Study of IMC-A12 in Patients With Thymoma and Thymic Carcinoma Who Have Been Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090212; 09-C-0212
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: Thymoma; Thymic Carcinoma; Thymic Carcinoid; Thymic Neuroendocrine Tumors
Keywords: Thymic Malignancies; IMC-A12; Insulin-Like Growth Factor
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thymoma (Experimental): Patients will receive IMC-A12 at a dose of 20 mg/kg intravenously once every three weeks. The most common tumors of the thymus are thymomas (well differentiated neoplasms and moderately differentiated neoplasms) and thymic (poorly differentiated neoplasms) carcinomas.
  Interventions: Drug: IMC-12
- Thymic Carcinoma (Experimental): Patients will receive IMC-A12 at a dose of 20 mg/kg intravenously once every three weeks. The most common tumors of the thymus are thymomas (well differentiated neoplasms and moderately differentiated neoplasms) and thymic (poorly differentiated neoplasms) carcinomas.
  Interventions: Drug: IMC-12

INTERVENTIONS:
Drug: IMC-12 — 20 mg/kg intravenously once every three weeks

SUMMARY:
Background:

* Cisplatin-containing chemotherapy is the standard of care for advanced thymoma and thymic carcinoma that cannot be treated with surgery. New options for treatment are necessary in patients with advanced thymoma and thymic carcinoma that have progressed on cisplatin-containing therapy.
* IMC-A12 is a new (experimental) agent that has not yet been approved by the Food and Drug Administration. IMC-A12 blocks the Insulin-like Growth Factor 1 receptor (IGF-1R). IGF-1R is found on many types of cancer cells, including cancer of the thymus, and is thought to play an important role in helping these cells to grow and divide.

Objectives:

* To determine if IMC-A12 has an effect on tumor growth in patients with cancer of the thymus.
* To evaluate the safety and tolerability of IMC-A12 in treatment for cancer of the thymus.

Eligibility:

- Individuals older than 18 years of age who have cancer of the thymus (thymoma, thymic carcinoma, or thymic carcinoid tumors) that has progressed in spite of standard treatment.

Design:

* Treatment will take place in 21-day cycles. Patients will receive one dose of IMC-A12 intravenously once every 3 weeks at the Clinical Center. During the Clinical Center visits, researchers will perform study tests and procedures to see how the study drugs are affecting the body.
* Patients will undergo a number of tests and procedures during the treatment cycle, including physical examinations, blood and urine samples for standard tests, imaging studies (ultrasound, magnetic resonance imaging (MRI) or computed tomography (CT) scans) to evaluate tumor growth, and blood and urine samples to evaluate the amount of IMC-A12 in the body.
* Patients may continue to take the drug as long as there are no adverse side effects and as long as the tumor does not grow.

DETAILED DESCRIPTION:
Background:

Cisplatin-containing chemotherapy is the standard of care for advanced unresectable thymoma and thymic carcinoma. New options for treatment are necessary in patients with advanced thymoma and thymic carcinoma that have progressed on cisplatin-containing therapy. The insulin-like growth factor (IGF) pathway is being studies in various malignancies including thymoma and thymic carcinoma. IMCA12 is an anti-IGF-1R monoclonal antibody that has shown activity in patients with thymic malignancies.

Objectives:

* To determine the objective response rate (partial response (PR)+complete response (CR)) to IMC-A12 monotherapy in patients with advanced or recurrent thymoma or thymic carcinoma.
* To evaluate time to response, duration of response, progression-free survival (PFS) and overall survival (OS)
* To assess safety of IMC-A12
* To perform immunohistochemistry for IGF1R expression on tumor samples of thymoma and thymic carcinoma (exploratory)
* To correlate response to therapy with changes in fludeoxyglucose 18F-positron emission tomography (FDG-PET) imaging at baseline and first restaging
* To perform pharmacokinetic (PK) analysis of IMC-A12
* To perform pharmacodynamic (PD) analysis in blood for the detection of IGF1R, AKT and pAKT in peripheral blood mononuclear cells (PBMC's) (exploratory).
* To assess circulating endothelial cell, circulating endothelial progenitor cells, immune subset analysis and glucose transport in peripheral blood monocytes and lymphocytes (exploratory).
* To evaluate anti-cytokine antibodies in peripheral blood (exploratory).

Eligibility:

* Patients with histologically confirmed thymic carcinoma or thymoma who have previously been treated on at least one platinum-containing chemotherapy regimen
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Adequate renal, hepatic and hematopoietic function
* No major surgery, radiotherapy, chemotherapy or biologic therapy within 28 days of IMC-A12 therapy

Design:

* Patients will receive IMC-A12 at a dose of 20 mg/kg intravenously once every three weeks
* Treatment with IMC-A12 alone will continue until disease progression
* Toxicity will be assessed every cycle by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 until December 31, 2010, and by CTCAE Version 4.0 beginning January 1, 2011
* Tumor response assessments by RECIST 1.0 criteria will be performed every 2 cycles
* Correlative studies including tissue immunohistochemistry studies will be done on existing tumor blocks
* Blood samples will be collected for for PK's, PD's, circulating endothelial cells (CEC's), circulating endothelial precursor cells (CEPC's), immune subsets, glucose transport and cytokine antibodies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically confirmation of invasive recurrent or metastatic thymoma or thymic carcinoma by the pathology department / Center for Cancer Research (CCR) / National Cancer Institute (NCI), or the pathology department of participating institutions.
* Patients must have had at least one prior platinum-containing chemotherapy regimen. There is no limit to the number of prior chemotherapy regimens received. Progressive disease should have been documented before entry into the study.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than 20 mm with conventional techniques or as greater than 10 mm with spiral CT scan. See section 11 for the evaluation of measurable disease.
* Target lesions cannot be selected within previously irradiated areas, if not newly arising or clearly progressing after irradiation as proven by repeat scanning.
* Patients must have recovered from toxicity related to prior therapy to at least to grade 1 (defined by CTCAE 3.0 until December 31, 2010, and by CTCAE 4.0 beginning January 1, 2011) and must not have had major surgery, radiation therapy, chemotherapy, biologic therapy (including any investigational agents), or hormonal therapy (other than replacement), within 4 weeks prior to entering the study.
* Concurrent corticosteroids for myasthenia gravis, or other paraneoplastic syndromes which often accompany thymic malignancies are allowed. Inhaled steroids are also allowed. However since steroids might occasionally induce responses in thymic malignancies patients should be on a stable dose of steroids for greater than or equal to 8 weeks before enrollment in order not to confound the efficacy assessment.
* Age greater than 18 years. Because no dosing or adverse event data are currently available on the use of IMC-A12 in patients less than 16 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials.
* Life expectancy of greater than 3 months.
* Performance status Eastern Cooperative Oncology Group (ECOG) less than or equal to 2.
* Patients must have adequate organ and marrow function (as defined below). Patients must have returned to baseline or grade 1 from any acute toxicity related to prior therapy:

  * leukocytes greater than or equal to 3,000/mm^3
  * absolute neutrophil count greater than or equal to 1,500/mm^3
  * hemoglobin greater than or equal to 9 g/dL
  * platelets greater than or equal to 100,000/mm^3
  * total bilirubin less than or equal to 1.5 times the institutional upper limit of normal (ULN)
  * aspartate aminotransferase (AST)(SGOT)/alanine aminotransferase (ALT)(SGPT) less than or equal to 3 times the institutional ULN

    (5x if LFT elevations due to liver metastases)
  * creatinine less than or equal to 1.5 times the institutional ULN

OR

--creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal

* Patients may be transfused to obtain a hemoglobin of 9.0.
* The patient must have fasting serum glucose less than 120 mg/dL or below the institutional ULN
* The effects of IMC-A12 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study therapy and for 3 months after the last dose of IMC-A12. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to comply with intravenous administration schedule, and the ability to understand and the willingness to sign a written informed consent document.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women and members of all races and ethnic groups are eligible for this trial. Every effort will be made to recruit women and minorities in this study.

EXCLUSION CRITERIA:

* Patients with symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 3 months without steroids may be enrolled at the discretion of the principal investigator.
* Patients with poorly controlled diabetes mellitus. Patients with a history of diabetes mellitus are allowed to participate, provided their blood glucose is within the normal range (fasting less than 120 mg/dL or below institutional upper limit of normal) and if they are on a stable dietary or therapeutic regimen for this condition.
* Uncontrolled medical illness including, but not limited to, ongoing or uncontrolled, symptomatic congestive heart failure (American Heart Association (AHA) Class II or worse), uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Human Immunodeficiency virus (HIV) positive patients with poorly controlled viral loads (viral load greater than 50 copies HIV/ml), and/or AIDS-defining illnesses will be excluded due to the possibility that IMC-A12 may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to IMC-A12. HIV positive patients with thymic malignancies not meeting the above criteria can be considered for inclusion in the study.
* Patients may not be receiving any other investigational agents.
* History of another invasive malignancy in the last five years. Adequately treated non-invasive, non-melanoma skin cancers, in situ carcinoma of the cervix, and surgically-removed papillary thyroid cancer will be allowed.
* Prior treatment with drugs of the IGF-1R inhibitor class.
* Patients with tumor amenable to potentially curative therapy as assessed by the investigator.
* Pregnant women are excluded from this study because IMC-A12 is a monoclonal antibody to IGF-1R with the potential for teratogenic or abortifacient effects. IgG antibody may also potentially be secreted in milk and therefore breastfeeding women should be excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IMC-A12.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-08; Primary Completion 2012-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giaccone G, Wilmink H, Paul MA, van der Valk P. Systemic treatment of malignant thymoma: a decade experience at a single institution. Am J Clin Oncol. 2006 Aug;29(4):336-44. doi: 10.1097/01.coc.0000227481.36109.e7. PMID 16891859
- [Background] Giaccone G. Treatment of malignant thymoma. Curr Opin Oncol. 2005 Mar;17(2):140-6. doi: 10.1097/01.cco.0000152628.43867.8e. PMID 15725919
- [Background] Okumura M, Ohta M, Tateyama H, Nakagawa K, Matsumura A, Maeda H, Tada H, Eimoto T, Matsuda H, Masaoka A. The World Health Organization histologic classification system reflects the oncologic behavior of thymoma: a clinical study of 273 patients. Cancer. 2002 Feb 1;94(3):624-32. doi: 10.1002/cncr.10226. PMID 11857293
- [Result] Rajan A, Carter CA, Berman A, Cao L, Kelly RJ, Thomas A, Khozin S, Chavez AL, Bergagnini I, Scepura B, Szabo E, Lee MJ, Trepel JB, Browne SK, Rosen LB, Yu Y, Steinberg SM, Chen HX, Riely GJ, Giaccone G. Cixutumumab for patients with recurrent or refractory advanced thymic epithelial tumours: a multicentre, open-label, phase 2 trial. Lancet Oncol. 2014 Feb;15(2):191-200. doi: 10.1016/S1470-2045(13)70596-5. Epub 2014 Jan 15. PMID 24439931
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0212.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The thymic carcinoma cohort was closed after enrolment of 12 participants because of lack of activity.
Period: Overall Study
Arm/Group | Thymoma | Thymic Carcinoma
Started | 37 | 12
Completed | 37 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thymoma | Thymic Carcinoma | Total
Number analyzed (Participants) | 37 | 12 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 11 | 39
  >=65 years | 9 | 1 | 10
Gender [Count of Participants; unit: Participants]
  Female | 18 | 5 | 23
  Male | 19 | 7 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 25 | 5 | 30
  White, Hispanic | 2 | 1 | 3
  Black | 6 | 1 | 7
  Asian | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 37 | 12 | 49
Median age [Median (Full Range); unit: years] | 52 [31 to 86] | 55 [26 to 71] | 52 [26 to 86]
Metastatic Sites [Number; unit: participants] — Data on metastatic sites is provided for 41 patients (29 thymoma, 12 thymic carcinoma) enrolled at the NCI. Eight thymoma patients were enrolled at Memorial Sloan Kettering Cancer Center, New York.
  participants
    Intrathoracic sites only | 18 | 0 | 18
    Extrathoracic sites(w/without intrathoracic sites | 11 | 12 | 23
Histological Analysis (WHO classification) [Number; unit: participants] — WHO (World Health Organization) classification of epithelial thymic malignancies: AB - Mixed, B1 - Predominantly cortical thymoma, B2 - Cortical thymoma, B2/B3 - Cortical thymoma/Well differentiated thymoma, B3 - Well differentiated thymoma, and C - Thymic carcinoma.
  participants
    AB | 2 | 0 | 2
    B1 | 4 | 0 | 4
    B2 | 15 | 0 | 15
    B2/B3 | 3 | 0 | 3
    B3 | 9 | 0 | 9
    C | 0 | 12 | 12
    Not otherwise specified | 4 | 0 | 4
Paraneoplastic Syndromes [Number; unit: participants]
  Myastenia gravis | 9 | 0 | 9
  Shulman's syndrome | 1 | 0 | 1
  Pure red-cell aplasia | 3 | 0 | 3
  Crohn's disease | 1 | 0 | 1
  Ulcerative colitis | 1 | 0 | 1
  Mucocutaneous candidiasis | 1 | 0 | 1
Previous systemic treatment (number of regimens) [Median (Full Range); unit: regimens] | 3 [1 to 11] | 2 [1 to 11] | 2 [1 to 11]
Previous systemic treatment (six or more regimens) [Number; unit: participants] | 10 | 2 | 12
Previous chemotherapy [Number; unit: participants]
  One line | 12 | 7 | 19
  Two lines | 8 | 2 | 10
  Three or more lines | 17 | 3 | 20
Previous platinum treatment [Number; unit: participants] | 37 | 12 | 49
Previous anthracycline [Number; unit: participants] | 27 | 5 | 32
Investigational drugs [Number; unit: participants] — Counted as previous lines of systemic treatment, but not as previous lines of chemotherapy.
  participants | 17 | 4 | 21
Previous radiotherapy [Number; unit: participants] | 23 | 4 | 27
Previous surgery [Number; unit: participants]
  Radical | 28 | 2 | 30
  Debulking | 1 | 1 | 2
  Biopsy | 8 | 9 | 17
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants]
  0 - Normal Activity | 3 | 1 | 4
  1 - Symptoms, but ambulatory | 29 | 8 | 37
  2 - In bed <50% of the time | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Partial Response (PR)+Complete Response (CR)) to IMC-A12 Monotherapy in Patients With Advanced or Recurrent Thymoma or Thymic Carcinoma.
Description: Objective response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response (CR) is the disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Patients were assessed for response every 2 cycles (every 6 weeks) while receiving the study drug.
Measure: Number; unit: Participants
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 37 | 12
Participants
  Complete Response | 0 | 0
  Partial Response | 5 | 0
  Stable Disease | 28 | 5
  Progressive Disease | 4 | 7

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 81 months and 17 days
Population: Adverse events are not separated by group because the adverse events are related to the drug which was the same in both groups.
Measure: Number; unit: Participants
Groups:
- IMC-A12 Monotherapy in Patients: Patients will receive IMC-A12 at a dose of 20 mg/kg intravenously once every three weeks.
Arm/Group | IMC-A12 Monotherapy in Patients
Number analyzed (Participants) | 49
Participants | 49

3. Secondary Outcome: Percentage of Participants Who Respond to Treatment
Description: Percentage of participants who respond to treatment was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: 39 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 37 | 12
percentage of participants | 14 [5 to 29] | 0 [0 to 26]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate is defined as objective response plus stable disease.
Time Frame: 39 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 37 | 12
percentage of participants | 89 [75 to 97] | 42 [15 to 72]

5. Secondary Outcome: Time to Progression
Description: Time between the first day of treatment to the day of disease progression.
Time Frame: 39 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 37 | 12
Months | 9.9 [7.3 to 12.8] | 1.7 [0.9 to 2.7]
Statistical Analysis 1: Comparison: Thymoma vs Thymic Carcinoma; Test type: Superiority or Other; p < 0.0001, Kaplan Meier

6. Secondary Outcome: Overall Survival
Description: Time from treatment start date until date of death or date last known alive.
Time Frame: 39 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 37 | 12
Months | 27.5 [15.0 to NA] — NA represents an undefined upper limit of the confidence interval because there were insufficient events (deaths) for it to be determined. | 8.4 [4.7 to 12.8]
Statistical Analysis 1: Comparison: Thymoma vs Thymic Carcinoma; Test type: Superiority or Other; p < 0.0001, Kaplan Meier

7. Secondary Outcome: Median Number of Cycles of Therapy
Description: A cycle is defined as 21 days or 6 weeks of therapy.
Time Frame: 6 weeks
Measure: Median (Full Range); unit: Cycles
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 37 | 12
Cycles | 13 [2 to 46] | 2.5 [1 to 8]

8. Secondary Outcome: Correlate Response to Therapy With Changes in FDG-PET Imaging
Description: Participants with scans that showed neither sufficient shrinkage to qualify as an objective response nor sufficient increase to qualify as disease progression, taking as reference the smallest cumulative longest dimension since start of treatment, to have stable disease.
Time Frame: 6 weeks after initiation of treatment
Population: We did radiological assessment ourselves, and an independent radiological assessment was not undertaken for assessment of response or progression.
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events are not separated by group because the adverse events are related to the drug which was the same in both groups.
Arm/Group | IMC-A12 Monotherapy in Patients
Serious Adverse Events (participants affected / at risk) | 29/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 Monotherapy in Patients (N=49)
Death NOS (General disorders) | 22 (22)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
CPK increased (Metabolism and nutrition disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Enterocolitis infection (Infections and infestations) | 1 (1)
Fever (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial infection (Cardiac disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mailgnant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — (not incl cysts and polyps) - Other, specify
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 Monotherapy in Patients (N=49)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 7 (12)
Acute coronary syndrome (Cardiac disorders) | 2 (2)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 23 (60)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 17 (31)
Allergic reaction (Immune system disorders) | 2 (2)
Allergic rhinitis (Immune system disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 35 (105)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (31)
Diarrhea (Gastrointestinal disorders) | 9 (22)
Dizziness (Nervous system disorders) | 5 (8)
Dry eye (Eye disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Dysgeusia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (20)
Ear and labyrinth disorders - Other, specify (patient reports of diminished hearing) (Ear and labyrinth disorders) | 1 (1)
Edema: limbs (Blood and lymphatic system disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3)
Eye disorders - Other, specify (Aur; lost vision R eye) (Eye disorders) | 2 (2)
Eye pain (Eye disorders) | 1 (1)
Fatigue (General disorders) | 18 (44)
Fever (General disorders) | 3 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flashing lights (Eye disorders) | 3 (3)
Floaters (Eye disorders) | 4 (5)
Flu like symptoms (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (5) — Oral ulcer; oral sensitivity; swallowing
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (11)
Hearing impaired (Ear and labyrinth disorders) | 3 (4)
Hemorroids (Gastrointestinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 14 (26)
Hyperglycemia (Metabolism and nutrition disorders) | 37 (182)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (24)
Hypermagnesemia (Metabolism and nutrition disorders) | 9 (20)
Hypernatremia (Metabolism and nutrition disorders) | 10 (17)
Hyperuricemia (Metabolism and nutrition disorders) | 22 (57)
Hypoalbuminemia (Metabolism and nutrition disorders) | 39 (110)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (20)
Hypoglycemia (Metabolism and nutrition disorders) | 7 (10)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 20 (59)
Hypotension (Cardiac disorders) | 2 (2)
INR increased (Blood and lymphatic system disorders) | 1 (1)
Infections and infestations - Other, specify (Opportunistic; thrush) (Infections and infestations) | 2 (2)
Infusion related reaction (Immune system disorders) | 1 (1)
Insomnia (General disorders) | 2 (2)
Investigations-Other, specify (Bicarbonate, serum-low) (Investigations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lipase increased (Metabolism and nutrition disorders) | 6 (22)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (3)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 20 (63)
lymphocyte count increased (Blood and lymphatic system disorders) | 8 (14)
Mucosal infection (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 9 (18)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder-Other, specify (Musculoskeletal and connective tissue disorders) | 13 (15) — Cramps; cramps lower extremity; hand cramps; hands cramps; hands, feet; leg cramps
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 17 (27)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mailgnant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — (incl cysts and polyps)-Other, specify (progression)
Neutrophil count decreased (Blood and lymphatic system disorders) | 8 (29)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Oral pain (Gastrointestinal disorders) | 2 (3)
Pain (General disorders) | 3 (6)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (12)
Platelet count decreased (Blood and lymphatic system disorders) | 16 (45)
Postnasal drip (Immune system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - Other, specify (urinary hesitancy) (Renal and urinary disorders) | 1 (1)
Serum amylase increased (Metabolism and nutrition disorders) | 8 (18)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4) — Brittle nails; hives; nail splitting
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Tumor pain (General disorders) | 8 (11)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Urinary tract infection (Renal and urinary disorders) | 4 (4)
Vertigo (Nervous system disorders) | 5 (8)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (18)
Weight loss (General disorders) | 6 (14)
White blood cell decreased (Blood and lymphatic system disorders) | 11 (40)
Hyponatremia (Metabolism and nutrition disorders) | 30 (78)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Metabolism and nutrition disorders) | 17 (68)
Constipation (Gastrointestinal disorders) | 7 (16)
Anorexia (Gastrointestinal disorders) | 20 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 23 (59)
Ataxia (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder infection (Infections and infestations) | 3 (3)
Bronchopulmonary hemorrhage (Blood and lymphatic system disorders) | 3 (4)
CPK increased (Metabolism and nutrition disorders) | 9 (17)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Metabolism and nutrition disorders) | 8 (26)
Blurred vision (Eye disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 6 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 (11)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2)
Facial muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No